CLINICAL TRIAL: NCT05754957
Title: A Phase 3, Randomized, Double-blind, Placebo-controlled, Event-driven Study to Demonstrate the Efficacy and Safety of Milvexian, an Oral Factor XIa Inhibitor, After a Recent Acute Coronary Syndrome
Brief Title: A Study of Milvexian in Participants After a Recent Acute Coronary Syndrome
Acronym: LIBREXIA-ACS
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR109271; 70033093ACS3003 (Other: Janssen Research & Development, LLC); 2022-501418-69-00 (Registry Identifier: EUCT number)
Record Dates: First submitted 2023-02-23; First posted 2023-03-06 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Acute Coronary Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — milvexian

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Milvexian (Experimental): Participants enrolled within 7 days of an acute coronary syndrome (ACS), who have undergone cardiac catheterization with percutaneous intervention (PCI) or who are being managed conservatively with or without catheterization, and who are receiving antiplatelet therapy standard-of-care (single antiplatelet therapy [SAPT] or dual antiplatelet therapy [DAPT]) as determined by the investigator will receive milvexian 25 milligrams (mg), orally, twice daily.
  Interventions: Drug: Milvexian
- Placebo (Placebo Comparator): Participants enrolled within 7 days of an ACS, who have undergone cardiac catheterization with PCI or who are being managed conservatively with or without catheterization, and who are receiving antiplatelet therapy standard-of-care (SAPT or DAPT) as determined by the investigator will receive placebo orally, twice daily.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Milvexian — Milvexian will be administered orally.
  Other Names: JNJ-70033093; BMS-986177
  Arms: Milvexian
Other: Placebo — Placebo will be administered orally.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate that milvexian is superior to placebo, in addition to standard-of-care, in reducing the risk of major adverse cardiovascular event (MACE) (the composite of cardiovascular [CV] death, myocardial infarction [MI], and ischemic stroke).

ELIGIBILITY:
Inclusion Criteria:

* Participants must have an index event that meets all 3 of the following criteria within 7 days prior to randomization: a) clinical syndrome consistent with spontaneous cardiac ischemia, b) diagnosis of acute coronary syndrome (ACS) (that is, ST-elevation myocardial infarction [STEMI], non-STEMI, or unstable angina [UA]), c) cardiac biomarker elevation (example, troponin I, troponin T, creatine kinase-MB [CK-MB]) above the upper limit of normal as determined by the local laboratory
* Participants must have at least 2 of the following risk factors:a) age 65 or older, b) diabetes mellitus, c) history of a prior myocardial infarction (MI) (other than index ACS event), d) multivessel coronary artery disease (CAD), e) history of coronary artery bypass graft (CABG) surgery prior to index ACS event, f) history of peripheral artery disease (PAD) or cerebrovascular disease (example, carotid atherosclerosis, intracranial artery stenosis, g) conservative management (that is, no percutaneous intervention [PCI] or CABG after index ACS event), h) Any one or more of the following high-risk angiographic features i) total stent length of greater than (>) 30 millimeters (mm), ii) thrombotic target lesion, iii) bifurcation lesion treated with more than one stent, iv) calcified target lesion treated with atherectomy, v) treatment of obstructive left main or proximal left anterior descending artery for index ACS (or clinical diagnosis of an anterior STEMI)
* All female participants of childbearing potential must have a negative highly sensitive serum beta-human chorionic gonadotropin (hCG) or urine test at screening
* A female participant must not be pregnant, breastfeeding, or planning to become pregnant until 4 days (5 half-lives) after the last dose of study intervention

Exclusion Criteria:

* MI secondary to ischemia due to either increased oxygen demand or decreased supply (Type 2 MI) or periprocedural MI as the index ACS event
* Planned CABG or staged PCI after randomization
* Any condition that requires chronic anticoagulation at the discretion of the investigator and/or local guidelines
* Conditions with a significant increased risk of bleeding (example, clinically significant bleeding within previous 3 months, known bleeding diathesis, et cetera)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14194 (Actual)
Dates: Start 2023-04-07 (Actual); Primary Completion 2026-09-07 (Estimated); Study Completion 2026-10-19 (Estimated)

PRIMARY OUTCOMES:
Time to First Occurrence of Major Adverse Cardiovascular Event (MACE) | Up to 3 years 6 months
  Time to first occurrence of any component of MACE will be reported. MACE is a composite of cardiovascular (CV) death, myocardial infarction (MI), and ischemic stroke.

SECONDARY OUTCOMES:
Time to the First Occurrence of Major Adverse Vascular Event (MAVE) | Up to 3 years 6 months
  Time to first occurrence of any component of MAVE will be reported. MAVE is a composite of CV death, MI, ischemic stroke, major adverse limb event (MALE), and symptomatic venous thromboembolism (VTE).
Time to the First Occurrence of Composite of All-cause Mortality (ACM), Myocardial Infarction (MI) and Ischemic Stroke | Up to 3 years 6 months
  Time to the first occurrence of composite of ACM, MI and ischemic stroke will be reported.
Time to Cardiovascular (CV) Death | Up to 3 years 6 months
  Time to CV death will be reported.
Time to All-cause Mortality (ACM) | Up to 3 years 6 months
  Time to ACM will reported. ACM will be categorized into CV death, non-CV death, and death due to unknown cause.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (997):
- United States (162):
  - Advanced Cardiovascular, LLC, Alexander City, Alabama
  - SORRA Research, Birmingham, Alabama
  - Ascension St. Vincent's Health System, Birmingham, Alabama
  - IMC-Diagnostic and Medical Clinic, Mobile, Alabama
  - Cardiology Associates of Mobile Inc, Mobile, Alabama
  - Mercy Gilbert Medical Center, Gilbert, Arizona
  - Valleywise Health Medical Center, Phoenix, Arizona
  - HonorHealth Neurology, Scottsdale, Arizona
  - Arkansas Heart Hospital, Little Rock, Arkansas
  - Bakersfield Memorial Hospital, Bakersfield, California
  - Mission Cardiovascular Research Institute, Fremont, California
  - Radin Cardiovascular Medical Group, Newport Beach, California
  - Valley Clinical Trials, Inc., Northridge, California
  - Stanford University School of Medicine, Palo Alto, California
  - VA Palo Alto Healthcare System, Palo Alto, California
  - Huntington Hospital, Pasadena, California
  - The Cardiovascular Center, Redding, California
  - University Of California San Diego, San Diego, California
  - San Diego Cardiac Center, San Diego, California
  - VA San Diego Health Care System, San Diego, California
  - UCLA, Santa Monica, California
  - NorthBay Clinical Research, LLC, Santa Rosa, California
  - Ramin Manshadi, MD, Stockton, California
  - South Denver Cardiology Associates PC, Littleton, Colorado
  - Nuvance Health Medical Practices Cardiology Danbury, Danbury, Connecticut
  - Cardiology Associates of Fairfield County, P.C., Stamford, Connecticut
  - George Washington University Medical Center, Washington D.C., District of Columbia
  - FWD Clinical Research, Boca Raton, Florida
  - Clearwater Cardiovascular Consultants, Clearwater, Florida
  - Holy Cross Hospital Inc., Fort Lauderdale, Florida
  - Integrative Research Associates, Fort Lauderdale, Florida
  - University of Florida Health Jacksonville, Gainesville, Florida
  - Inpatient Research Clinic LLC, Hialeah, Florida
  - Shands Jacksonville Medical Center Inc dba UF Health Jacksonville, Jacksonville, Florida
  - Cardiology Partners Clinical Research Institute, Loxahatchee Groves, Florida
  - Baptist Hospital of Miami, Miami, Florida
  - Advanced Research for Health Improvement, Naples, Florida
  - Amavita Clinical Research (Dr. Pedro Martinez-Clark), North Miami Beach, Florida
  - South Florida Research Solutions LLC, Pembroke Pines, Florida
  - Coastal Cardiology Consultants, Safety Harbor, Florida
  - Cardiovascular Center of Sarasota, Sarasota, Florida
  - Tampa Cardiovascular Interventions and Research, Tampa, Florida
  - Interventional Cardiac Consultants, Trinity, Florida
  - Cardiology Partners Clinical Research Institute, Wellington, Florida
  - Grady Memorial Hospital, Atlanta, Georgia
  - Atlanta Clinical Research Center, Cartersville, Georgia
  - Northeast Georgia Heart Center, Gainesville, Georgia
  - Cardiovascular Consultants of South Georgia LLC, Thomasville, Georgia
  - Kootenai Medical Center, Coeur d'Alene, Idaho
  - Insight Hospital and Medical Center Chicago, Chicago, Illinois
  - Illinois Heart and Vascular Foundation, Chicago, Illinois
  - Advocate Heart Institute, Downers Grove, Illinois
  - Clinical Investigation Specialists, Inc., Gurnee, Illinois
  - Essential Concepts Research Solutions, Palos Hills, Illinois
  - OSF HealthCare Cardiovascular Institute, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Prairie Cardiovascular Consultants, Ltd., Springfield, Illinois
  - Carle Foundation Hospital, Urbana, Illinois
  - Midwest Cardiovascular Research Foundation, Elkhart, Indiana
  - Northern Indiana Research Alliance, Fort Wayne, Indiana
  - IU Health Ball Memorial Hospital, Muncie, Indiana
  - Reid Health, Richmond, Indiana
  - Health Midwest Ventures Group, Inc d b a HCA MidAmerica Division, LLC, Overland Park, Kansas
  - University of Louisville, Louisville, Kentucky
  - Norton Cardiovascular Associates, Louisville, Kentucky
  - Cambridge Medical Trials, Alexandria, Louisiana
  - Cardiovascular Institute of the South, Houma, Louisiana
  - Ochsner Clinic And Hospital, New Orleans, Louisiana
  - Louisiana Heart Center, Slidell, Louisiana
  - Monroe Research LLC, West Monroe, Louisiana
  - Eastern Maine Medical Center Northeast Cardiology Associates, Bangor, Maine
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - Suburban Hospital, Bethesda, Maryland
  - Captiol Cardiology Associates, Lanham, Maryland
  - Shady Grove Office, Rockville, Maryland
  - Tidal Health Peninsula Regional Inc., Salisbury, Maryland
  - Pentucket Medical Associates, Haverhill, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - St. Joseph Mercy Oakland, Bloomfield Hills, Michigan
  - AAMRC, Flint, Michigan
  - Jackson Heart Clinic, Jackson, Michigan
  - Sparrow Clinical Research Institute, Lansing, Michigan
  - St. Luke's Cardiology Associates, Duluth, Minnesota
  - HealthEast Medical Research Institute, Saint Paul, Minnesota
  - Mercy Medical Research Institute, Chesterfield, Missouri
  - The Curators of the University of Missouri on behalf of University of Missouri Health Care, Columbia, Missouri
  - North Kansas City Hospital, Kansas City, Missouri
  - Spectrum Clinical Research, Kansas City, Missouri
  - Cox Health, Springfield, Missouri
  - Saint Louis University, St Louis, Missouri
  - Bryan LGH Heart Institute, Lincoln, Nebraska
  - Methodist Physicians Clinic Heart Consultants, Omaha, Nebraska
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Ash Research Clinic, Brick, New Jersey
  - Englewood Health, Englewood, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Atlanticare Regional Medical Center, Pomona, New Jersey
  - Cardio Metabolic Institute, Somerset, New Jersey
  - Buffalo General Medical Center, Buffalo, New York
  - Jamaica Hospital Medical Center, Jamaica, New York
  - Columbia University Medical Center, New York, New York
  - Weil Cornell University, New York, New York
  - Weill Cornell Medicine, New York, New York
  - Hudson Valley Cardiovascular Practice, PC, Poughkeepsie, New York
  - Cardiac Care & Vascular Medicine, PLLC, The Bronx, New York
  - Westchester Medical Center, Valhalla, New York
  - Clinical Trials of America, Cary, North Carolina
  - UNC School of Medicine, Chapel Hill, North Carolina
  - The Moses H. Cone Memorial Hospital, Greensboro, North Carolina
  - Atrium Health Wake Forest Baptist, High Point, North Carolina
  - Clinical Trials of America, Lenoir, North Carolina
  - Novant Health, Matthews, North Carolina
  - Rex Hospital, Raleigh, North Carolina
  - Sanford Cardiology, Sanford, North Carolina
  - Trinity Medical Group, Minot, North Dakota
  - Summa Health System, Akron, Ohio
  - University of Cincinnati, Cincinnati, Ohio
  - Metro Health Hospital, Cleveland, Ohio
  - Ohio Health, Columbus, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - The Heart House, Springfield, Ohio
  - Ascension Medical Group - St. John Clinic Infectious Disease, Bartlesville, Oklahoma
  - South Oklahoma Heart Research, Oklahoma City, Oklahoma
  - St John Health System Inc, Tulsa, Oklahoma
  - Advanced Cardiac Care, Bethlehem, Pennsylvania
  - Chambersburg Hospital, Chambersburg, Pennsylvania
  - Hamot Medical Center, Erie, Pennsylvania
  - UPMC Pinnacle Health, Harrisburg, Pennsylvania
  - St. Mary Medical Center, Langhorne, Pennsylvania
  - Penn Presbyterian Medical Center, Philadelphia, Pennsylvania
  - Lankenau Institute for Medical Research, Wynnewood, Pennsylvania
  - AnMed Health, Anderson, South Carolina
  - Prisma Health, Greenville, South Carolina
  - St. Francis Physician Services, Inc, DBA Upstate Cardiology Research, Greenville, South Carolina
  - Carolina Cardiology Associates, Rock Hill, South Carolina
  - Monument Health Clinical Research, Rapid City, South Dakota
  - Erlanger Health System, Chattanooga, Tennessee
  - Apex Cardiology, Jackson, Tennessee
  - Ascension Saint Thomas West Hospital, Nashville, Tennessee
  - Vanderbilt University, Nashville, Tennessee
  - Parkway Cardiology Associates PC, Oak Ridge, Tennessee
  - Amarillo Heart Clinical Research Institute, Amarillo, Texas
  - PharmaTex Research, Amarillo, Texas
  - Med Research, Inc., El Paso, Texas
  - Texas Tech University Health Sciences Center-El Paso, El Paso, Texas
  - Baylor Scott and White Research Institute, Fort Worth, Texas
  - East Texas Cardiology, PA, Houston, Texas
  - Physician Research Network, Houston, Texas
  - Vital Heart and Vein, Humble, Texas
  - Texas Cardiology Research Center, Kingwood, Texas
  - Ascension Texas Cardiovascular, Kyle, Texas
  - Cardiovoyage, Sherman, Texas
  - Northwest Heart Clinical Research, LLC., Tomball, Texas
  - Virginia Heart, Falls Church, Virginia
  - Riverside Regional Medical Center, Newport News, Virginia
  - Sentara Cardiovascular Research Institute, Norfolk, Virginia
  - Winchester Medical Center, Winchester, Virginia
  - Providence Regional Medical Center Everett, Everett, Washington
  - Cardiac Surgery Group, Tacoma, Washington
  - MultiCare Health System, Tacoma, Washington
  - Mayo Clinic Health System, La Crosse, Wisconsin
  - Marshfield Clinic, Marshfield, Wisconsin
- Argentina (40):
  - Hospital Espanol De Bahia Blanca, Bahía Blanca
  - Hospital Italiano Regional Del Sur, Bahía Blanca
  - Hospital Italiano de Buenos Aires, Buenos Aires
  - Sanatorio Finochietto, Buenos Aires
  - Hospital Britanico de Buenos Aires, Buenos Aires
  - Sanatorio Guemes, CABA
  - Centro Medico Dra. Laura Maffei - Investigacion Clinica Aplicada, Ciudad Autonoma Buenos Aires
  - Instituto Cardiovascular de Buenos Aires, Ciudad Autonoma Buenos Aires
  - Fundacion Favaloro, Ciudad Autonoma Buenos Aires
  - Clinica Adventista Belgrano, Ciudad Autonoma Buenos Aires
  - Clinica Coronel Suarez, Coronel Suárez
  - Clínica Chutro, Córdoba
  - Hospital San Roque, Córdoba
  - Sanatorio Duarte Quiroz, Córdoba
  - Clinica Romagosa, Córdoba
  - Clinica Privada del Prado, Córdoba
  - Sanatorio Allende, Córdoba
  - Sanatorio de la Canada, Córdoba
  - Instituto Privado De Especialidades Medicas S.A. Fundacion J Robert Cade, Córdoba
  - Hospital Cordoba, Córdoba
  - Centro Medico Luquez, Córdoba
  - Hospital Privado Centro Medico de Cordoba, Córdoba
  - Hospital Italiano de La Plata, La Plata
  - Centro de Investigaciones Medicas Mar Del Plata, Mar del Plata
  - Sanatorio Modelo de Quilmes, Quilmes
  - Instituto Cardiovascular de Rosario, Rosario
  - Sanatorio Parque, Rosario
  - Hospital Italiano Garibaldi, Rosario
  - Hospital Provincial del Centenario, Rosario
  - Centro de Investigaciones Clinicas Salta, Salta
  - Centro Cardiovascular Salta, Salta
  - Hospital El Cruce, San Juan Bautista
  - Corporacion Medica de Gral. San Martin S.A., San Martín
  - Investigaciones Clinicas Tucuman, San Miguel de Tucumán
  - Estudios Clinicos de los Arroyos, San Nicolás
  - Sanatorio Mayo SA, Santa Fe
  - Hospital José María Cullen, Santa Fe
  - Sanatorio Medico de Diagnostico y Tratamiento, Santa Fe
  - Sanatorio San Martin, Venado Tuerto
  - Clinica Privada Fusavim SRL, Villa María
- Australia (18):
  - Royal Adelaide Hospital, Adelaide
  - Flinders Medical Centre, Adelaide
  - Ballarat Base Hospital, Ballarat
  - Sunshine Coast University Hospital, Birtinya
  - Cairns Base Hospital, Cairns
  - Royal Prince Alfred Hospital, Camperdown
  - Concord Repatriation General Hospital, Concord
  - The Canberra Hospital, Garran
  - Royal Brisbane and Women's Hospital, Herston
  - Royal Hobart Hospital, Hobart
  - Nepean Hospital, Kingswood
  - Core Research Group, Milton
  - Fiona Stanley Hospital, Murdoch
  - Gold Coast University Hospital, Southport
  - Westmead Hospital, Sydney
  - Latrobe Regional Hospital, Traralgon
  - Wollongong Hospital, Wollongong
  - The Queen Elizabeth Hospital, Woodville South
- Austria (5):
  - KH St.Josef Braunau am Inn, Braunau am Inn
  - Landeskrankenhaus Feldkirch, Feldkirch
  - LKH-Univ. Klinikum Graz, Graz
  - Krankenhaus der Elisabethinen Linz, Linz
  - AKH - Medizinische Universitat Wien, Vienna
- Belgium (16):
  - Imeldaziekenhuis, Bonheiden
  - AZ Klina, Brasschaat
  - AZ Sint-Jan, Bruges
  - C.H.U. Brugmann, Brussels
  - CUB Hôpital Erasme, Brussels
  - Universitair Ziekenhuis Brussel, Brussels
  - Cliniques Universitaires Saint Luc, Brussels
  - Ziekenhuis Oost-Limburg, Genk
  - AZ Sint-Lucas, Ghent
  - Jessa Ziekenhuis, Hasselt
  - CHR de la Citadelle, Liège
  - Az Sint-Maarten, Mechelen
  - Heilig Hart Ziekenhuis Lier, Mol
  - CHU Ambroise Pare, Mons
  - AZ Delta, Roeselare
  - AZ Turnhout, Turnhout
- Brazil (52):
  - Hospital Vera Cruz, Belo Horizonte
  - IMINC Instituto Mineiro de Intervencao Cardiologica LTDA, Belo Horizonte
  - Cardresearch - Cardiologia Assistencial, Belo Horizonte
  - Instituto das Pequenas Missionárias de Maria Imaculada - Hospital Madre Teresa, Belo Horizonte
  - UNESP - Faculdade de Medicina da Universidade Estadual Paulista - Campus Botucatu, Botucatu
  - Hospital do Coracao do Brasil, Brasília
  - Centro de Cardiologia Clinica e Pesquisa Doutora Juliana Souza Ltda CECAP Centro de Cardiologia Clinica, Brasília
  - Sociedade Hospitalar Angelina Caron, Campina Grande do Sul
  - C.E.C.-Centro Especializado em Cardiologia Ltda.- Loema Medicina e Bem Estar, Campinas
  - Instituto de Pesquisa Clinica de Campinas, Campinas
  - Sociedade Literaria e Caritativa Santo Agostinho Hospital Sao Jose, Criciúma
  - Irmandade Santa Casa de Misericordia de Curitiba, Curitiba
  - Associacao Paranaense de Cultura PUCPR, Curitiba
  - Hospital Cardiológico Costantini, Curitiba
  - Hospital Das Clinicas Da Universidade Federal De Goias, Goiânia
  - Instituto do Coracao de Marília, Marília
  - Instituto Atena de Pesquisa Clinica, Natal
  - Instituto Mederi de Pesquisa e Saude, Passo Fundo
  - Santa Casa de Misericordia de Pelotas, Pelotas
  - Hospital Maternidade e Pronto Socorro Santa Lucia, Poços de Caldas
  - Associacao Hospitalar Moinhos de Vento, Porto Alegre
  - Hospital das Clinicas de Porto Alegre, Porto Alegre
  - IMV Pesquisa Cardiologica Sociedade Simples HMD COR l, Porto Alegre
  - Hospital Ernesto Dornelles, Porto Alegre
  - Uniao Brasileira de Educacao e Assistencia Hospital Sao Lucas da PUCRS, Porto Alegre
  - Fundacao Universitaria de Cardiologia, Porto Alegre
  - Hospital Nossa Senhora da Conceicao S A, Porto Alegre
  - PROCAPE - Universidade de Pernambuco Pronto Socorro Cardiológico de Pernambuco prof Luiz Tavares, Recife
  - Secretaria de Saude Hospital Agamenon Magalhaes, Recife
  - Hospital Das Clinicas Da Faculdade De Medicina De RPUSP HCRP, Ribeirão Preto
  - Hospital sao lucas, Rio de Janeiro
  - Hospital Santa Izabel Santa Casa de Misericordia da Bahia, Salvador
  - Instituto CardioPulmonar, Salvador
  - Fundacao Bahiana de Cardiologia, Salvador
  - Hospital da Bahia, Salvador
  - Pesquisare Saude, Santo André
  - CEMEC - Centro Multidisciplinar de Estudos Clínicos, São Bernardo do Campo
  - Instituto de Cardiologia de Santa Catarina, São José
  - Fundacao Faculdade Regional de Medicina de Sao Jose do Rio Preto Hospital de Base, São José do Rio Preto
  - Irmandade Da Santa Casa De Misericordia De Sao Paulo, São Paulo
  - FGM Clinica Paulista de Doencas Cardiovasculares Ltda, São Paulo
  - Real e Benemerita Associacao Portuguesa de Beneficencia, São Paulo
  - Hospital Alemao Oswaldo Cruz, São Paulo
  - Instituto Dante Pazzanese de Cardiologia, São Paulo
  - Hospital Das Clinicas Da Faculdade De Medicina Da USP, São Paulo
  - Sociedade Beneficente Israelita Brasileira Hospital Albert Einstein, São Paulo
  - Casa de Saude Santa Marcelina - Hospital Santa Marcelina, São Paulo
  - Instituto de Moléstias Cardiovasculares Tatuí, Tatuí
  - HC-UFTM - Hospital de Clínicas da Universidade Federal do Triângulo Mineiro, Uberaba
  - Clinica Cardioped Ltda, Vitória
  - CEDOES, Vitória
  - Santa Casa de Misericórdia de Votuporanga, Votuporanga
- Bulgaria (19):
  - MHAT Puls, Blagoevgrad
  - MHAT Heart and Brain, Burgas
  - Multiprofile Hospital for Active Treatment Dr. Tota Venkova, Gabrovo
  - Multiprofile Hospital for Active Treatment - Haskovo, Haskovo
  - MHAT Uni Hospital, Panagyurishte
  - SHATC Sveti Georgi-Pernik OOD, Pernik
  - Multiprofile Hospital for Active Treatment Heart and Brain, Pleven, Pleven
  - UMHAT 'Dr. Georgi Stranski', EAD, Pleven
  - UMHAT 'Sv. Georgi' EAD, Plovdiv
  - MHAT Sv. Karidad EAD, Plovdiv
  - 2th MHAT - Sofia, Sofia
  - National Heart Hospital, Sofia
  - Diagnostic Consultation Centre 'Alexandrovska' EOOD, Sofia
  - UMHAT Prof. Dr. Aleksandar Chirkov, Sofia
  - University Multiprofile Hospital for Active Treatment - Tsaritsa Yoanna - ISUL, EAD, Sofia
  - UMHATEM N I Pirogov, Sofia
  - University Multiprofile Hospital for Active Treatment- UMHAT Sveta Anna AD, Sofia
  - UMHAT Sofia Med, Sofia
  - UMHAT Prof. Dr. St. Kirkovich AD, Stara Zagora
- Canada (26):
  - Foothills Hospital, Calgary, Alberta
  - University of Alberta, Edmonton, Alberta
  - Surrey Memorial Hospital, Surrey, British Columbia
  - Vancouver General Hospital, Vancouver, British Columbia
  - Saint Boniface General Hospital, Winnipeg, Manitoba
  - Dalhousie University, Halifax, Nova Scotia
  - Dr. Saul Vizel Cardiac Research Office, Cambridge, Ontario
  - Hamilton Health Sciences Corporation, Hamilton, Ontario
  - London Health Sciences Centre, London, Ontario
  - Southlake Regional Health Centre, Newmarket, Ontario
  - Halton Healthcare Services Corporation, Oakville, Ontario
  - University of Ottawa Heart Institute, Ottawa, Ontario
  - Kawartha Cardiology Clinical Trials, Peterborough, Ontario
  - Niagara Health System, St. Catharines, Ontario
  - Toronto Sunnybrook Hospital, Toronto, Ontario
  - Office of Dr. Anthony Glanz, Windsor, Ontario
  - Clinique de Cardiologie de Levis, Lévis, Quebec
  - Centre de Recherche du CHUM, Montreal, Quebec
  - Montreal General Hospital, Montreal, Quebec
  - Montreal Heart Institute, Québec, Quebec
  - Centre de Recherche Clinique de Quebec, Québec, Quebec
  - Institut Universitaire De Cardiologie Et De Pneumologie De Québec, Québec, Quebec
  - CardioVasc HR, Saint-Jean-sur-Richelieu, Quebec
  - CSSS du Sud de Lanaudiere - Hopital Pierre-Le Gardeur d/b/a CISSS de Lanaudiere, Terrebonne, Quebec
  - CIUSSS de la Mauricie-et-du-Centre-du-Quebec, Trois-Rivières, Quebec
  - Royal University Hospital, Saskatoon, Saskatchewan
- Chile (5):
  - Quantum Research, Puerto Varas
  - Centro de Investigacion Clinica Universidad Catolica de Chile CICUC, Santiago
  - Centro de Estudios Cardiologicos y de Medicina Interna, Temuco
  - Centro de Investigacion Clinica del Sur, Temuco
  - Centro de Estudios Clinicos V Region Ltda, Viña del Mar
- China (61):
  - Baotou Central Hospital, Baotou
  - Beijing Anzhen Hospital, Capital Medical University, Beijing
  - Peking University First Hospital, Beijing
  - Beijing Shijitan Hospital, Beijing
  - Beijing Friendship Hospital Capital Medical University, Beijing
  - Peking University Third Hospital, Beijing
  - Chinese PLA General Hospital, Beijing
  - The First Hospital of Jilin University, Changchun
  - Changzhou No 2 Peoples Hospital, Changzhou
  - West China Hospital Sichuan University, Chengdu
  - Sichuan Provincial Peoples Hospital, Chengdu
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing
  - Dongguan People s Hospital, Dongguan
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou
  - Guangdong Provincial People's Hospital, Guangzhou
  - The First Affiliated Hospital of Sun Yat-Sen University, Guangzhou
  - The Affiliated Hospital of Guizhou Medical University, Guiyang
  - GuiZhou Privicial Peoples Hospital, Guiyang
  - Zhejiang Provincial People's Hospital, Hangzhou
  - Affiliated Hangzhou First People's Hospital, Zhejiang University School of Medicine, Hangzhou
  - Sir Run Run Shaw Hospital Zhejiang University School of Medicine, Hangzhou
  - Anhui Province Hospital, Hefei
  - Huizhou Municipal Central Hospital, Huizhou
  - Qilu Hospital of Shandong University, Jinan
  - The Second Affiliated Hospital, Shandong University, Jinan
  - Shandong Jining No.1 People's Hospital, Jining
  - Lanzhou University Second Hospital, Lanzhou
  - Linfen Central Hospital, Linfen
  - The Second Affiliated Hospital of Nanchang University, Nanchang
  - Nanjing Drum Tower Hospital, Nanjing
  - Zhongda Hospital Southeast University, Nanjing
  - Jiangsu Province Hospital, Nanjing
  - The First Affiliated Hospital of Nanyang Medical College, Nanyang
  - Ningbo First Hospital, Ningbo
  - Shanghai Ninth Peoples Hospital, Shanghai
  - Shanghai Chest Hospital, Shanghai
  - Zhongshan Hospital Fudan University, Shanghai
  - The First Affiliated Hospital of Shantou University Medical, Shantou
  - Fuwai Hospital Chinese Academy of Medical Sciences, Shenzhen, Shenzhen
  - The Second Affiliatted Hospital of Soochow University, Suzhou
  - The First Affiliated Hospital of Soochow University, Suzhou
  - Shanxi Cardiovascular Hospital, Taiyuan
  - Tianjin Medical University General Hospital, Tianjin
  - Tianjin People's Hospital, Tianjin
  - The Second Hospital Of Tianjin Medical University, Tianjin
  - Tianjin Chest Hospital, Tianjin
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou
  - Wenzhou Peoples Hospital, Wenzhou
  - The Central Hospital of Wuhan, Wuhan
  - Hubei Zhongshan Hospital The Third Peoples Hospital of Hubei Province, Wuhan
  - Wuxi People s Hospital, Wuxi
  - The First Affiliated Hospital of Xian Jiaotong University, Xi'an
  - The Third Affiliated Hospital of Xinxiang Medical University, Xinxiang
  - The Affiliated Hospital of Xuzhou Medical College, Xuzhou
  - Yanbian University Hospital, Yanji
  - Yichang Central Pepole's Hospital, Yichang
  - General Hospital of Ningxia Medical Hospital, Yinchuan
  - Affiliated Hospital Of Guangdong Medical University, Zhanjiang
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou
  - Zhongshan City Peoples Hospital, Zhongshan
  - Affiliated Hospital of Zunyi Medical University, Zunyi
- Croatia (6):
  - General Hospital Dubrovnik, Dubrovnik
  - Special Hospital for medical rehabilitation, Krapinske Toplice
  - Clinical Hospital Centre Rijeka, Rijeka
  - General Hospital Slavonski Brod, Slavonski Brod
  - Poliklinika Solmed, Zagreb
  - University Hospital Dubrava, Zagreb
- Czechia (18):
  - Fakultni nemocnice Brno, Brno
  - Vojenska nemocnice Brno, Brno
  - Fakultni nemocnice u sv. Anny v Brne, Brno
  - Nemocnice Ceske Budejovice a s, České Budějovice
  - Fakultni nemocnice Hradec Kralove, Hradec Králové
  - Kardiocentrum Vysocina CZ a.s., Jihlava
  - Oblastní nemocnice Kolín, Kolín
  - Krajská nemocnice Liberec a.s., Liberec
  - Fakultni Nemocnice Ostrava, Ostrava-Poruba
  - Pardubicka krajska nemocnice a s, Pardubice
  - Fakultni nemocnice Plzen, Pilsen
  - Fakultni nemocnice Kralovske Vinohrady, Prague
  - Kardiologie Vinohrady s r o, Prague
  - Vseobecna fakultni nemocnice v Praze, Prague
  - Institut klinicke a experimentalni mediciny, Prague
  - Ustredni vojenske nemocnice Praha, Prague
  - Nemocnice Slany, Slaný
  - Nemocnice AGEL - Podlesi a.s., Třinec
- Denmark (9):
  - Aarhus University Hospital, Aahus N
  - Amager Hospital, Copenhagen S
  - Bispebjerg Og Frederiksberg Hospital, Frederiksberg
  - Herning Regional Hospital, Herning
  - Holbæk Sygehus, Holbæk
  - Hvidovre Hospital, Hvidovre
  - Slagelse Sygehus, Slagelse
  - Odense University Hospital, Svendborg
  - Viborg Hospital, Viborg
- France (30):
  - CHU Angers - Hopital Hotel Dieu, Angers
  - CH Prive Saint-Martin, Caen
  - CHRU de Tours - Hopital Trousseau, Chambray-lès-Tours
  - Centre Hospitalier Sud Francilien, Corbeil-Essonnes
  - Hopital Henri Mondor, Créteil
  - CHU Dijon, Dijon
  - CHU de Grenoble Hopital Albert Michallon, La Tronche
  - CH de Chartres - Hôpital Louis Pasteur, Le Coudray
  - CHRU de Lille Hopital Claude Huriez, Lille
  - Centre Hospitalier Saint Joseph Et Saint Luc, Lyon
  - Clinique Du Pont De Chaume, Montauban
  - CHU de Montpellier Hopital Saint Eloi, Montpellier
  - Centre Hospitalier Emile Muller, Mulhouse
  - CHU Nantes, Institut du thorax, Nantes
  - Centre Hospitalier Universitaire - de Nice - Hopital Pasteur, Nice
  - Hôpital Caremeau, Nîmes
  - Hopital Lariboisiere, Paris
  - Hopital Saint-Antoine, Paris
  - Hôpital Bichat - Claude Bernard, Paris
  - Hopital Cochin, Paris
  - Centre Hospitalier de Pau, Pau
  - Hôpital du Haut Lévêque, Pessac
  - CHU Poitiers - Hopital la Miletrie, Poitiers
  - Hopital de Bicetre, Potigny
  - CHU Rouen Hopital Charles Nicolle, Rouen
  - Clinique Saint-Hilaire - Centre Frédéric Joliot, Rouen
  - Nouvel Hopital Civil - CHU Strasbourg, Strasbourg
  - Hopital Rangueil, Toulouse
  - CHU de Nancy - Hopital de Brabois, Vandœuvre-lès-Nancy
  - Hopital Andre Mignot, Versailles
- Germany (35):
  - Klinikum am Plattenwald, Bad Friedrichshall
  - Universitaetsklinikum Freiburg, Bad Krozingen
  - Kerckhoff-Klinik Bad Nauheim, Bad Nauheim
  - Vivantes Klinikum Im Friedrichshain, Berlin
  - Charite Campus Benjamin Franklin, Berlin
  - Charité Campus Virchow, Berlin
  - Vivantes Humboldt Klinikum, Berlin
  - GFO Kliniken Bonn, Betriebsstaette St. Marien, Beuel
  - Klinikum Bielefeld, Bielefeld
  - Marienhausklinikum Eifel Bitburg, Bitburg
  - Universitatsklinikum Bonn, Bonn
  - Staedisches Klinikum Brandenburg, Brandenburg
  - Hospital Bremen Mitte, Bremen
  - Regiomed Klinikum Coburg, Coburg
  - St. Johannes-Hospital, Dortmund
  - Staedtisches Klinikum Dresden Standort Dresden Friedrichstadt, Dresden
  - Katholisches Krankenhaus St. Josef gGmbH - Abtlg. für Gynäkologie, Erfurt
  - Klinikum der Johann Wolfgang Goethe -Universitaet, Frankfurt
  - Universitaetsmedizin Greifswald, Greifswald
  - Universitaetsklinikum Hamburg Eppendorf, Hamburg
  - Asklepios Klinik Barmbek, Hamburg
  - Asklepios Klinik St. Georg, Hamburg
  - Klinikum Leverkusen gGmbH, Leverkusen
  - Herzzentrum Ludwigshafen, Ludwigshafen
  - Klinikum Luedenscheid, Lüdenscheid
  - Universitätsklinikum Magdeburg, Magdeburg
  - Katholisches Klinikum Mainz; Innere Medizin I- Kardiologie, Mainz
  - Universitatsmedizin der Johannes Gutenberg Universitat Mainz, Mainz
  - Universitaetsklinikum Mannheim, Mannheim
  - Kliniken Maria Hilf GmbH, Mönchengladbach
  - Marienhaus Klinikum, Neuwied
  - Sana-Klinikum Remscheid GmbH, Remscheid
  - Universitaetsmedizin Rostock, Rostock
  - Universitaetsklinikum Tuebingen, Tübingen
  - Klinikum Worms gGmbH, Worms
- Greece (16):
  - Uni General Hospital of Alexandroupolis, Alexandroupoli
  - Henry Dunant Hospital, Athens
  - General Hospital of Athens G Gennimatas, Athens
  - Hippokration Hospital, Athens
  - General Hospital of Athens Attikon, Athens
  - General Hospital of Attiki 'KAT', Athens
  - Athens Medical Center, Athens
  - General Per Hospital of Athens Asklipiio Voulas, Athens
  - University Hospital of Heraklion, Heraklion
  - University General Hospital of Ioannina, Ioannina
  - University Hospital Of Larissa, Larissa
  - General University Hospital of Patras, Pátrai
  - Ahepa University General Hospital of Thessaloniki, Thessaloniki
  - Hippokration Hospital, Thessaloniki
  - Papageorgiou General Hospital, Thessaloniki
  - Papanikolaou General Hospital of Thessaloniki, Thessaloniki
- Hungary (15):
  - Budai Irgalmasrendi Korhaz, Budapest
  - Semmelweis Egyetem, Budapest
  - Gottsegen György Országos Kardiológiai Intézet, Budapest
  - Bajcsy-Zsilinszky Kórház és Rendelőintézet, Budapest
  - Semmelweis Egyetem Varosmajor Sziv es Ergyogyaszati Klinika, Budapest
  - Debreceni Egyetem, Debrecen
  - Bekes Megyei Kozponti Korhaz Pandy Kalman Tagkorhaz, Gyula
  - Somogy Megyei Kaposi Mor Oktato Korhaz, Kaposvár
  - Bacs-kiskun Megyei Korhaz, Kecskemét
  - Pecsi Tudomanyegyetem, Pécs
  - Szegedi Tudományegyetem Áok Szent-Györgyi Albert Klinikai Központ, Szeged
  - Tolna Megyei Balassa Janos Korhaz, Szekszárd
  - Jasz Nagykun Szolnok Megyei Hetenyi Geza Korhaz Rendelointez, Szolnok
  - Markusovszky Egyetemi Oktatokorhaz, Szombathely
  - Belvarosi Egeszseghaz Kft. (Leda-Platan Maganklinika es Sebeszeti Kozpont), Zalaegerszeg
- India (29):
  - NHL Medical College (SVP Hospital IMSR), Ahmedabad
  - Jawaharlal Nehru Medical College and Hospital, Aligarh
  - Sri Jayadeva Institute, Bangalore
  - KLE's Dr. Prabhakar Kore Hospital & Medical Research Centre (MRC), Belagavi
  - S.P.Medical College & AG of Hospitals, Bikaner
  - Tamil Nadu Government Multi Super Speciality Hospital, Chennai
  - Apollo Hospitals, Chennai
  - Batra Hospital And Medical Research Centre, Delhi
  - Osmania General Hospital, Hyderabad
  - Care Hospitals, Hyderbad
  - Lisie Hospital, Kochi
  - NRS Medical College, Kolkata
  - IPGMER and SSKM Hospital, Kolkata
  - Rabindranath Tagore International Institute of Cardiac Sciences, Kolkata
  - Dayanand Medical College & Hospital, Tagore Nagar, Civil Lines, Ludhiana
  - Kasturba Medical College Hospital, Mangalore
  - Seth G S Medical College and KEM Hospital, Mumbai
  - Arneja Heart Institute, Nagpur
  - Crescent Hospital & Heart Center, Nagpur
  - Central India Cardiology Hospital and Research Institute, Nagpur
  - All India Institute of Medical Sciences, New Delhi
  - Sir Ganga Ram Hospital, New Delhi
  - Indira Gandhi Institute of Medical Sciences, Patna
  - Ruby Hall Clinic, Pune
  - KEM Hospital & Research Centre, Pune
  - Nanjappa Hospital, Shimoga
  - Unicare Heart Institute, Surat
  - Government Siddhartha Medical College, Vijayawada
  - King George Hospital, Visakhapatnam
- Israel (19):
  - Haemek Medical Center, Afula
  - Samson Assuta Ashdod University Hospital, Ashdod
  - Barzilai Medical Center, Ashkelon
  - Soroka University Medical Center, Beersheba
  - Bnai Zion Medical Center, Haifa
  - Rambam Health Care Campus, Haifa
  - Carmel Medical Center, Haifa
  - Wolfson Medical Center, Holon
  - Shaare Zedek Medical Center, Jerusalem
  - Hadassah University Hospita Ein Kerem, Jerusalem
  - Hadassah Medical Center, Jerusalem
  - Meir Medical Center, Kfar Saba
  - Health Corporation of Galilee Medical Center, Naharya
  - Rabin Medical Center, Petah Tikva
  - Chaim Sheba Medical Center, Ramat Gan
  - Kaplan Medical Center, Rehovot
  - Assaf Harofeh Medical Center, Rishon LeZiyyon
  - Ziv Medical Center, Safed
  - Baruch Padeh Medical Center, Tiberias
- Italy (23):
  - Azienda Ospedaliera Nazionale SS. Antonio e Biagio e Cesare Arrigo Alessandria, Alessandria
  - Cliniche Humanitas Gavazzeni, Bergamo
  - Azienda Socio Sanitaria Territoriale Papa Giovanni XXIII (Presidio Papa Giovanni XXIII), Bergamo
  - Azienda USL di Bologna - Ospedale Maggiore, Bologna
  - Universita D Annunzio, Chieti
  - Azienda Ospedaliero-Universitaria di Ferrara Arcispedale Sant Anna, Ferrara
  - Ospedale Sant'Andrea, La Spezia
  - Azienda Ulss 3 Serenissima distretto di Mirano, Mestre
  - Fondazione IRCCS Ca Granda Ospedale Maggiore Policlinico, Milan
  - Centro Cardiologico Monzino, Milan
  - Azienda Socio Sanitaria Territoriale Niguarda (Grande Ospedale Metropolitano Niguarda), Milan
  - Azienda Ospedaliera Universitaria Federico II, Napoli
  - Azienda Ospedaliero Universitaria di Parma, Parma
  - Fondazione IRCCS Policlinico San Matteo, Pavia
  - A. O.U. Pisana Ospedale di Cisanello, Pisa
  - AOU Policlinico Umberto I, Roma
  - Fondazione Policlinico Universitario A Gemelli IRCCS, Roma
  - Istituto Clinico Humanitas, Rozzano
  - Ospedale San Francesco, Sassari
  - Ospedale Bolognini, Seriate
  - IRCCS Multimedica di Sesto San Giovanni, Sesto San Giovanni
  - Azienda Ospedaliero Universitaria Ospedali Riuniti, Torrette Di Ancona
  - Azienda Ospedaliera Ospedale Treviglio-Caravaggio di Treviglio, Treviglio
- Japan (71):
  - Kasugai Municipal Hospital, Aichi
  - Hyogo Prefectural Amagasaki General Medical Center, Amagasaki Shi
  - Chiba University Hospital, Chiba
  - Funabashi Municipal Medical Center, Chiba
  - Saiseikai Futsukaichi Hospital, Chikushino-shi
  - Fukui Prefectural Hospital, Fukui-shi
  - National Hospital Organization Kyushu Medical Center, Fukuoka
  - Fukuoka Wajiro Hospital, Fukuoka
  - Kyushu University Hospital, Fukuoka
  - Gifu Prefectural General Medical Center, Gifu
  - National Hospital Organization Takasaki General Medical Center, Gunma
  - Hyogo Prefectural Harima-Himeji General Medical Center, Himeji-shi
  - Hiratsuka Kyosai Hospital, Hiratsuka-shi
  - Hirosaki University Hospital, Hirosaki
  - Hiroshima City Hiroshima Citizens Hospital, Hiroshima
  - Tokai University Hospital, Isehara
  - Public Central Hospital of Matto Ishikawa, Ishikawa
  - Teikyo University Hospital, Itabashi Ku
  - Juntendo University Shizuoka Hospital, Izunokuni-shi
  - Tesshokai Kameda Clinic, Kamogawa
  - Showa University Fujigaoka Hospital, Kanagawa
  - Asanokawa, Kanazawa Cardiovascular Hospital, Kanazawa
  - Fukuoka Tokushukai Hospital, Kasuga-shi
  - Kimitsu Chuo Hospital, Kisarazu-shi
  - Kokura Memorial Hospital, Kitakyushu-shi
  - Chikamori Hospital, Kochi
  - National Hospital Organization Fukuoka Higashi Medical Center, Koga
  - Kumamoto University Hospital, Kumamoto
  - Saiseikai Kumamoto Hospital, Kumamoto
  - Kurashiki Central Hospital, Kurashiki
  - National Hospital Organization Kure Medical Center and Chugoku Cancer Center, Kure-shi
  - Kyoto University Hospital, Kyoto
  - National Hospital Organization Kyoto Medical Center, Kyoto
  - Tokushukai Chiba-Nishi General Hospital, Matsudo-shi
  - Jisenkai Aizawa Hospital, Matsumoto-shi
  - Toho University Medical Center, Ohashi Hospital, Meguro-ku
  - Tokyo Saiseikai Central Hospital, Minatoku
  - Miyazaki Medical Association Hospital, Miyazaki
  - NHO Nagoya Medical Center, Nagoya
  - Japanese Red Cross Aichi Medical Center Nagoya Daini Hospital, Nagoya
  - Hyogo Medical University Hospital, Nishinomiya Shi
  - Okayama Rosai Hospital, Okayama
  - Osaka City General Hospital, Osaka
  - National Hospital Organization Osaka National Hospital, Osaka
  - Osaka Police Hospital, Osaka
  - Saga University Hospital, Saga
  - Kitasato University Hospital, Sagamihara
  - National Hospital Organization Saitama National Hospital, Saitama
  - Iwatsuki Minami Hospital, Saitama-shi
  - Tohoku University Hospital, Sendai
  - Showa University Hospital, Shinagawa City
  - Tokyo Women's Medical University Hospital, Shinjuku-ku
  - Iwate Medical University Hospital, Shiwa-gun
  - National Cerebral and Cardiovascular Center, Suita-Shi
  - Kagawa Prefectural Central Hospital, Takamatsu
  - Tokushima University Hospital, Tokushima
  - Mitsui Memorial Hospital, Tokyo
  - St. Luke's International Hospital, Tokyo
  - Nippon Medical School Hospital, Tokyo
  - National Hospital Organization Tokyo Medical Center, Tokyo
  - Nihon University Itabashi Hospital, Tokyo
  - Ome Medical Center, Tokyo
  - Toyama Prefectural Central Hospital, Toyama
  - Mie University Hospital, Tsu
  - Tsuchiura Kyodo General Hospital, Tsuchiura
  - Tsukuba Medical Center Hospital, Tsukuba
  - Yamaguchi University Hospital, Ube
  - Tokyo Bay Urayasu Ichikawa Medical Center, Urayasu-shi
  - National Hospital Organization Ureshino Medical Center, Ureshino-shi
  - Wakayama Medical University Hospital, Wakayama
  - Yokohama City University Medical Center, Yokohama
- Latvia (3):
  - Daugavpils Regional Hospital, Daugavpils
  - Riga East Clinical University Hospital, Riga
  - Pauls Stradins Clinical University Hospital, Riga
- Lithuania (3):
  - Hospital of Lithuanian University of Health Sciences Kaunas Clinics, Kaunas
  - Klaipeda Seamen's Hospital, Public Institution, Klaipėda
  - Vilnius University Hospital Santariskiu Clinic, Public Institution, Vilnius
- Malaysia (11):
  - Hospital University Sains Malaysia, Kota Bharu
  - Hospital Raja Perempuan Zainab Ii, Kota Bharu
  - Hospital Queen Elizabeth, Kota Kinabalu
  - Institut Jantung Negara, Kuala Lumpur
  - Pusat Perubatan Universiti Kebangsaan Malaysia, Kuala Lumpur
  - University Malaya Medical Centre, Kuala Lumpur
  - Sarawak General Hospital, Kuching
  - Hospital Miri, Miri
  - Hospital Pulau Pinang, Pulau Pinang
  - Hospital Seberang Jaya, Seberang Jaya
  - Universiti Teknologi Mara, Selayang Baru Utara
- Mexico (10):
  - Hospital Cardiologica Aguascalientes, Aguascalientes
  - Centro para el Desarrollo de la Medicina y de Asistencia Médica Especializada S.C., Culiacán
  - Centro de Estudios de de alta Especialidad de Sinaloa, Mazatlán
  - Instituto Nacional de Cardiologia Dr. Ignacio Chavez, México
  - Private Practice Dr Amaya, Monterrey
  - Centro de Estudios Clinicos de Queretaro S.C, Querétaro
  - Centro de Atencion e Investigacion Cardiovascular del Potosi S C, San Luis Potosí City
  - Centro de Investigacion Cardiovascular y Metabolica, Tijuana
  - Centro de Investigacion Dr. Alberto Esteban Bazzoni Ruiz, Torreón
  - Dr Enrique Lopez Rosas, Xalapa
- Netherlands (27):
  - Jeroen Bosch Ziekenhuis, 's-Hertogenbosch
  - Noordwest Ziekenhuisgroep, Alkmaar
  - Ziekenhuisgroep Twente, Almelo
  - Meander Medisch Centrum, Amersfoort
  - Onze Lieve Vrouwe Gasthuis, Amsterdam
  - Deventer Ziekenhuis, Deventer
  - Ziekenhuis Gelderse Vallei, Ede
  - Catharina Ziekenhuis, Eindhoven
  - Treant Zorggroep, Emmen
  - Medisch Spectrum Twente, Enschede
  - Admiraal De Ruyter Ziekenhuis - Goes, Goes
  - Groene Hart Ziekenhuis, Gouda
  - Ziekenhuis St Jansdal, Harderwijk
  - Zuyderland Medical Center, Heerlen
  - Elkerliek Ziekenhuis, Helmond
  - Alrijne Ziekenhuis Leiden ; Cardiology, Leiderdorp
  - Maastricht UMC, Maastricht
  - St. Antonius Ziekenhuis Nieuwegein, Nieuwegein
  - Radboudumc, Nijmegen
  - Bravis, Roosendaal
  - Sint Franciscus Gasthuis, Rotterdam
  - D & A Research, Sneek
  - Ziekenhuis Rivierenland, Tiel
  - Diakonessenhuis, Utrecht
  - Maxima Medisch Centrum, Veldhoven
  - VieCuri Medisch Centrum, Venlo
  - Gelre Ziekenhuizen Zutphen, Zutphen
- New Zealand (10):
  - North Shore Hospital, Auckland
  - Auckland City Hospital, Auckland
  - University of Otago, Christchurch
  - Dunedin Public Hospital, Dunedin
  - Hawkes Bay Hospital, Hastings
  - Taranaki Base Hospital, New Plymouth
  - Middlemore Hospital, Otahuhu
  - Rotorua Hospital, Rotorua
  - Tauranga Hospital, Tauranga
  - Whangarei Hospital, Whangarei
- North Macedonia (2):
  - University Clinic of Cardiology, Skopje
  - Clinical Hospital Tetovo, Tetovo
- Philippines (18):
  - The Heart Specialists Clinic and Diagnostic Center, Angeles
  - Silang Specialists Medical Center, Cavite
  - Cebu Doctors University Hospital, Cebu
  - Central Lab Diabetes Wellness, Heart and Kidneys, Inc, Davao City
  - Davao Doctors Hospital, Davao City
  - Southern Philippines Medical Center, Davao City
  - St.Paul's Hospital-Iloilo, Iloilo City
  - Mary Mediatrix Medical Center, Lipa City
  - Health Cube Medical Clinics, Mandaluyong
  - Manila Doctors Hospital, Manila
  - Medical Center Manila, Manila
  - Philippine General Hospital, Manila
  - Chinese General Hospital & Medical Center, Manila
  - Amang Rodriguez Memorial Medical Center, Marikina City
  - The Medical City, Pasig
  - St. Luke's Medical Center, Quezon
  - Cardinal Santos Medical Center, San Juan City
  - The Medical City South Luzon, Santa Rosa
- Poland (27):
  - Uniwersytecki Szpital Kliniczny w Bialymstoku, Bialystok
  - NZOZ Centrum Medyczne KERmed, Bydgoszcz
  - Samodzielny Publiczny Zaklad Opieki Zdrowotnej, Bytom
  - Wojewodzki Szpital Zespolony w Elblagu, Elblag
  - Clinical Medical Research Sp. z o.o., Katowice
  - Specjalistyczna Poradnia Kardiologiczna i Nadcisnienia Tetniczego, Kielce
  - Ewa Mirek-Bryniarska Specjalistyczna Praktyka Lekarska, Krakow
  - Krakowskie Centrum Kardiologii Inwazyjnej, Elektroterapii i Angiologii, Krakow
  - Krakowski Szpital Specjalistyczny im Jana Pawla II, Krakow
  - SPZOZ Centralny Szpital Kliniczny UM w Lodzi, Lodz
  - 1 Wojskowy Szpital Kliniczny Z Poliklinika SPZOZ W Lublinie, Lublin
  - Samodzielny Publiczny Szpital Kliniczny Nr 4 w Lublinie, Lublin
  - NZOZ Osrodek Kardiologii Inwazyjnej -Ikardia, Nałęczów
  - Wojewodzki Szpital Specjalistyczny w Olsztynie, Olsztyn
  - FutureMeds Olsztyn, Olsztyn
  - Medicome Sp. Z O.O., Oświęcim
  - Uniwersytet Medyczny im. Karola Marcinkowskiego w Poznaniu, Poznan
  - Wojewodzki Szpital im Sw Ojca Pio w Przemyslu, Przemyśl
  - Samodzielny Publiczny Szpital Wojewodzki im. Papieza Jana Pawla II, Siedlce
  - ETG Skierniewice, Skierniewice
  - NZOZ PRO CORDIS Sopockie Centrum Badan Kardiologicznych, Sopot
  - Wojewodzki Szpital Zespolony im L Rydygiera w Toruniu, Torun
  - Narodowy Instytut Kardiologii Stefana kardynala Wyszynskiego Panstwowy Instytut Badawczy, Warsaw
  - Specjalistyczny Szpital im dra Alfreda Sokolowskiego w Walbrzychu, Wałbrzych
  - Uniwersytecki Szpital Kliniczny im Jana Mikulicza Radeckiego we Wroclawiu, Wroclaw
  - 4 Wojskowy Szpital Kliniczny Z Poliklinika SP ZOZ, Wroclaw
  - Wojewodzki Szpital Specjalistyczny we Wroclawiu, Wroclaw
- Portugal (11):
  - Centro Hospitalar do Baixo Vouga E P E Unidade de Aveiro, Aveiro
  - Hospital de Braga, Braga
  - Uls Coimbra - Hosp. Univ. Coimbra, Coimbra
  - Centro Hospitalar Cova da Beira, EPE - Hospital Pêro da Covilhã, Covilha
  - Uls Alto Ave - Hosp. Sra. Da Oliveira Guimaraes, Guimarães
  - Centro Hospitalar de Leiria, Leiria
  - Centro Hospitalar de Lisboa Central, Lisbon
  - Centro Hospitalar de Lisboa Norte Hospital Santa Maria, Lisbon
  - Centro Hospitalar de Entre o Douro e Vouga, E.P.E, Santa Maria da Feira
  - Centro Hospitalar de Vila Nova de Gaia Espinho E P E, Vila Nova de Gaia
  - Centro Hospitalar de Trás os Montes e Alto Douro- Vila Real, Vila Real
- Romania (18):
  - Spitalul Judetean de Urgenta Dr. Constantin Opris, Baia Mare
  - Spitalul Clinic Judetean de Urgenta Brasov, Brasov
  - Spitalul Universitar de Urgenta Militar Central 'Dr. Carol Davila', Bucharest
  - Spitalul Universitar de Urgenta Elias, Clinica de Cardiologie, Bucharest
  - Spitalul Clinic de Urgenta Bucuresti, Bucharest
  - Institutul de urgenta pentru Boli Cardiovasculare Prof. Dr. C.C. Iliescu, Bucharest
  - Spitalul Angiocare SRL, Cluj-Napoca
  - Spitalul Clinic Judetean de Urgenta Cluj Napoca, Cluj-Napoca
  - Spitalul Clinic Judetean de Urgenta Sf. Apostol Andrei, Constanța
  - Spitalul Clinic Judetean de Urgenta Craiova, Craiova
  - Institutul de Boli Cardiovasculare Iasi, Iași
  - Spitalul Clinic Judetean de Urgenta Oradea, Oradea
  - SAL MED Pitesti, Piteşti
  - Spitalul Clinic Judetean de Urgenta Targu Mures, Târgu Mureş
  - Spitalul Clinic Judetean de Urgenta Targu Mures, Tg. Mures
  - Clinica Medicaliss, Timișoara
  - Spitalul Clinic Municipal de Urgenta Timisoara, Timișoara
  - Institutul de Boli Cardiovasculare Timisoara, Timișoara
- Serbia (14):
  - Clinical Center Dr Dragisa Misovic Dedinje, Belgrade
  - Institute for Cardiovascular diseases Dedinje, Belgrade
  - University Clinical Center of Serbia, Belgrade
  - Clinical Hospital Center Zemun, Belgrade
  - University Clinical Hospital Center Dr Dragisa Misovic- Dedi, Belgrade
  - Institute of Cardiovascular Diseases of Vojvodina, Kamenitz
  - University Clinical Center Kragujevac, Kragujevac
  - Clinical Center Nis, Niš
  - Institute for Treatment and Rehabilitation Niska Banja, Niška Banja
  - General Hospital Pancevo, Pančevo
  - General Hospital Smederevo, Smederevo
  - General Hospital Sremska Mitrovica, Sremska Mitrovica
  - General Hospital Uzice, Užice
  - Health Center Zajecar, Zaječar
- Singapore (5):
  - National University Hospital, Singapore
  - National Heart Centre (NHC) Singapore, Singapore
  - Changi General Hospital, Singapore
  - Ng Teng Fong General Hospital, Singapore
  - Khootech Puat Hospital, Singapore
- Slovakia (15):
  - Stredoslovensky ustav srdcovych a cievnych chorob a.s, Banská Bystrica
  - Alian s.r.o., Bardejov
  - Premedix Clinic, Bratislava
  - Nemocnica s poliklinikou Brezno, Brezno
  - Východoslovenský Ústav Srdcových A Cievnych Chorôb, A.S., Košice
  - Interno Kardio s r o, Košice
  - Kardiologicka ambulancia CARDIO D&R s.r.o., Košice
  - Kardio 1 S.R.O., Lučenec
  - Univerzitná nemocnica Martin, Martin
  - Kardiologicka ambulancia MEDI M&M s.r.o., Moldava nad Bodvou
  - Kardiocentrum Nitra s.r.o., Nitra
  - Cardioinvest s.r.o., Nové Zámky
  - Interna SK s.r.o., Svidník
  - Nemocnica AGEL Zvolen a s, Zvolen
  - MEDIVASA s.r.o., Žilina
- South Africa (11):
  - Panorama MediClinic, Cape Town
  - Tread Research, Cape Town
  - Tiervlei Trial Centre, Cape Town
  - Groote Schur Hospital, Cape Town
  - Johese Clinical Research, Centurion
  - Durban Medical Centre, Durban
  - Garda, RA, Johannesburg
  - Eden Heart, Mossel Bay
  - Dr J.M. Engelbrecht Trial Site, Somerset West
  - Helderberg Research Institute, Somerset West
  - Clinical Projects Research SA (PTY) LTD, Worcester
- South Korea (29):
  - Bucheon St. Mary's Hospital, Bucheon-si
  - Inje University Busan Paik Hospital, Busan
  - Pusan National University Hospital, Busan
  - Dong-A University Hospital, Busan
  - Chungbuk National University Hospital, Cheongju-si
  - Kangwon National University Hospital, Chuncheon
  - Keimyung University Dongsan Hospital, Daegu
  - Konyang University Hospital, Daejeon
  - Chungnam National University Hospital, Daejeon
  - Ewha Woman's University Seoul Hospital, Gangseo-gu
  - Myongji Hospital, Goyang-si
  - Chonnam National University Hospital, Gwangju
  - Seoul National University Bundang Hospital, Gyeonggi-do
  - Gachon University Gil Medical Center, Incheon
  - The Catholic University of Korea, Incheon St. Mary's Hospital, Incheon
  - Chungnam National University Sejong Hospital, Sejong-si
  - Korea University Anam Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - VHS Medical Center, Seoul
  - Asan Medical Center, Seoul
  - Gangnam Severance Hospital, Yonsei University Health System, Seoul
  - Seoul St.Mary s Hospital, Seoul
  - Severance Hospital Yonsei University Health System, Seoul
  - Kyung Hee University Hospital, Seoul
  - Kyung Hee University Hospital at Gangdong, Seoul
  - Hanyang University Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - WonJu Severance Christian Hospital, Wŏnju
  - Pusan National University Yangsan Hospital, Yangsan
- Spain (24):
  - Hosp. Gral. Univ. de Alicante, Alicante
  - Hosp. Del Mar, Barcelona
  - Hosp. de La Santa Creu I Sant Pau, Barcelona
  - Hosp Univ Vall D Hebron, Barcelona
  - Hosp Clinic de Barcelona, Barcelona
  - Hosp. Univ. Virgen de La Arrixaca, El Palmar
  - Hosp. de Cabuenes, Gijón
  - Hosp. Univ. Arnau de Vilanova de Lleida, Lleida
  - Hosp. Virgen de La Luz, Madrid
  - Hosp. Univ. de La Princesa, Madrid
  - Hosp. Univ. Ramon Y Cajal, Madrid
  - Hosp. Clinico San Carlos, Madrid
  - Hosp. Univ. 12 de Octubre, Madrid
  - Hosp. Univ. La Paz, Madrid
  - Hosp. Univ. Hm Monteprincipe, Madrid
  - Hosp. de Manises, Manises
  - Hosp Virgen de La Victoria, Málaga
  - Complejo Hosp. de Navarra, Pamplona
  - Hosp. Clinico Univ. de Santiago, Santiago de Compostela
  - Hosp. Univ. Joan Xxiii, Tarragona
  - Hosp. Clinico Univ. de Valencia, Valencia
  - Hosp. Gral. Univ. Valencia, Valencia
  - Hosp. Alvaro Cunqueiro, Vigo
  - Hosp. Univ. Miguel Servet, Zaragoza
- Switzerland (5):
  - Universitatsspital Basel, Basel
  - Universitätspital Bern, Universitätsklinik für Frauenheilkunde, Bern
  - Hopitaux Universitaires de Geneve - HUG, Geneva
  - Istituto Cardiocentro Ticino, Lugano
  - UniversitaetsSpital Zuerich, Zurich
- Taiwan (16):
  - Changhua Christian Hospital, Changhua
  - Kaohsiung Medical University Chung Ho Memorial Hospital, Kaohsiung City
  - E-DA Hospital, Kaohsiung City
  - Far Eastern Memorial Hospital, New Taipei City
  - Mackay Memorial Hospital, New Taipei City
  - China Medical University Hospital, Taichung
  - Chi Mei Medical Center Yong Kang, Tainan
  - National Taiwan University Hospital, Taipei
  - Cathay General Hospital, Taipei
  - Taipei Medical University, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Cheng Hsin General Hospital, Taipei
  - Tri-Service General Hospital, Taipei
  - Taipei Municipal Wanfang Hospital, Taipei
  - Chang Gung Memorial Hospital- Linkou, Taoyuan
  - National Yang-Ming University Hospital, Yilan County
- Thailand (5):
  - Ramathibodi Hospital, Bangkok
  - Siriraj Hospital, Bangkoknoi
  - Maharaj Nakorn Chiang Mai Hospital, Chiang Mai
  - Srinagarind Hospital, Nai Mueang Subdistrict Mueang
  - King Chulalongkorn Memorial Hospital, Pathum Wan
- Turkey (Türkiye) (14):
  - Afyon Kocatepe University Medical Faculty, Afyonkarahisar
  - Ankara Etlik Speciality Hospital, Ankara
  - Ankara University Medical Faculty, Ankara
  - Ankara Numune Research and Training Hospital, Ankara
  - Bursa Yuksek Ihtisas Training and Research Hospital, Bursa
  - Osmangazi University Medical Faculty, Eskişehir
  - Bezmi Alem Vakif University Medical Faculty Hospital, Istanbul
  - Marmara University Pendik Training Hospital, Istanbul
  - Dokuz Eylul University Medical Faculty, Izmir
  - Karabuk University Medical Faculty, Karabük
  - Erciyes University Medical Faculty, Kayseri
  - Kutahya Health Science University Evliya Celebi Research and Training Hospital, Kütahya
  - Mersin University Medical Faculty, Mersin
  - Ondokuz Mayis University, Samsun
- United Kingdom (35):
  - Basingstoke And North Hampshire Hospital, Basingstoke
  - Royal United Hospital, Bath
  - Queen Elizabeth Hospital, Birmingham
  - Birmingham Heartlands Hospital, Birmingham
  - Blackpool Victoria Hospital, Blackpool
  - Royal Bournemouth Hospital, Bournemouth
  - University Hospital Bristol and Weston NHS trust, Bristol
  - Dorset County Hospital, Dorchester
  - Russels Hall Hospital, Dudley
  - Hairmyres Hospital, East Kilbride
  - Royal Infirmary of Edinburgh, Edinburgh
  - Royal Devon and Exeter Hospital(Wonford), Exeter
  - Royal Free Hospital, Hampstead
  - Harefield Hospital, Harefield
  - West Middlesex University Hospital, Isleworth
  - Kingston Hospital, Kingston upon Thames
  - Leeds General Infirmary, Leeds
  - Lincoln County Hospital, Lincoln
  - Barts Hospital, London
  - Hammersmith Hospital, London
  - Altnagelvin Hospital, Londonderry
  - North Manchester General Hospital, Manchester
  - James Cook University Hospital, Middlesbrough
  - Freeman Hospital, Newcastle upon Tyne
  - Peterborough City Hospital, Peterborough
  - Derriford Hospital, Plymouth
  - Queen Alexandra Hospital, Portsmouth
  - East Surrey Hospital, Redhill
  - Lister Hospital, Stevenage
  - Morriston Hospital, Swansea
  - Musgrove Park Hospital, Taunton
  - Torbay Hospital-Devon, Torquay
  - Sandwell and West Birmingham Hospitals NHS Trust-Sandwell Gene, West Bromwich
  - Royal Albert Edward Infirmary, Wigan
  - Yeovil District Hospital, Yeovil
- Vietnam (9):
  - Bach Mai Hospital, Hanoi
  - Tam Anh General Hospital, Hanoi
  - 103 Military Hospital, Hanoi
  - Hanoi Heart Hospital, Hanoi
  - Hanoi Medical University Hospital, Hanoi
  - People's Hospital 115, Ho Chi Minh City
  - Tam Anh Hospital, Ho Chi Minh City
  - Thong Nhat HOSPITAL, Ho Chi Minh City
  - Tam Duc Heart Hospital, Ho Chi Minh City

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

REFERENCES:
- [Derived] Gibson CM, Bahit MC, Mehran R, Mehta SR, Lamee RA, Goto S, Weitz JI, Horrow J, Barnathan ES, Harrington RA, Mahaffey KW, Lam CSP, Pieper KS, Johnston SC, Hankey GJ, Plotnikov AN, Li D, Deng H, Steg PG; Librexia ACS Committees and Investigators.. Oral factor xia inhibitor milvexian after a recent acute coronary syndrome: Rationale and design of the phase 3 (Librexia ACS). Am Heart J. 2025 Jul;285:21-28. doi: 10.1016/j.ahj.2025.02.011. Epub 2025 Feb 20. PMID 39986336